CLINICAL TRIAL: NCT00666484
Title: Phase II Study Evaluating the Toxicity and Efficacy of a Modified German Paediatric Hodgkin's Lymphoma Protocol (HD95) in Young Adults (Aged 18-30 Years) With Hodgkin's Lymphoma
Brief Title: Combination Chemotherapy in Treating Younger Patients With Hodgkin Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000593560; UCL/07/005 (Other: University College London); 2007-003080-45 (EudraCT Number); EU-20844
Record Dates: First submitted 2008-04-24; First posted 2008-04-25 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Lymphoma; Neurotoxicity
Keywords: neurotoxicity; stage I adult Hodgkin lymphoma; stage II adult Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; adult lymphocyte depletion Hodgkin lymphoma; adult lymphocyte predominant Hodgkin lymphoma; adult mixed cellularity Hodgkin lymphoma; adult nodular sclerosis Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Neurotoxicity Syndromes; Hodgkin Disease | interventions — Cyclophosphamide; Doxorubicin; Etoposide; Prednisolone; Procarbazine; Vincristine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Treatment Group 1: stages 1A, 1B, 2A: OEPA x 2 (Experimental): OEPA (28day cycle):
  Vincristine 1.5mg/m^2 iv d1,d8,d15 (capped at 2mg/dose) Etoposide 125mg/m^2 iv d1-5 Prednisolone 60mg/m^2 po d1-15 Adriamycin 40mg/m^2 iv d1 and 15
  Interventions: Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: prednisolone; Drug: vincristine sulfate; Radiation: radiation therapy
- Treatment Group 2: stages 2AE, 2B, 3A: OEPA x 2 + COPP x 2 (Experimental): OEPA (28 day cycle) Vincristine 1.5mg/m^2 iv d1,d8,d15 (capped at 2mg/dose) Etoposide 125mg/m^2 iv d1-5 Prednisolone 60mg/m^2 po d1-15 Adriamycin 40mg/m^2 iv d1 and 15
  COPP (28 day cycle) Cyclophosphamide 500mg/m^2 iv d1 and 8 Vincristine 1.5mg/m^2 iv d1,8 (capped 2mg/dose) Procarbazine 100mg/m^2 po d1-15* Prednisolone 40mg/m^2 po d1-15
  Interventions: Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: prednisolone; Drug: procarbazine hydrochloride; Drug: vincristine sulfate; Radiation: radiation therapy
- Treatment Group 3: stages 2BE, 3AE, 3B, 4: OEPAx2 + COPPx4 (Experimental): OEPA (28 day cycle) Vincristine 1.5mg/m^2 iv d1,d8,d15 (capped at 2mg/dose) Etoposide 125mg/m^2 iv d1-5 Prednisolone 60mg/m^2 po d1-15 Adriamycin 40mg/m^2 iv d1 and 15
  COPP (28 day cycle) Cyclophosphamide 500mg/m^2 iv d1 and 8 Vincristine 1.5mg/m^2 iv d1,8 (capped 2mg/dose) Procarbazine 100mg/m^2 po d1-15* Prednisolone 40mg/m^2 po d1-15
  Interventions: Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: prednisolone; Drug: procarbazine hydrochloride; Drug: vincristine sulfate; Radiation: radiation therapy

INTERVENTIONS:
Drug: cyclophosphamide
  Arms: Treatment Group 2: stages 2AE, 2B, 3A: OEPA x 2 + COPP x 2; Treatment Group 3: stages 2BE, 3AE, 3B, 4: OEPAx2 + COPPx4
Drug: doxorubicin hydrochloride
Drug: etoposide
Drug: prednisolone
Drug: procarbazine hydrochloride
  Arms: Treatment Group 2: stages 2AE, 2B, 3A: OEPA x 2 + COPP x 2; Treatment Group 3: stages 2BE, 3AE, 3B, 4: OEPAx2 + COPPx4
Drug: vincristine sulfate
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. It is not yet known which regimen of combination chemotherapy is more effective for Hodgkin lymphoma.

PURPOSE: This phase II trial is studying the side effects of three different regimens of combination chemotherapy and to see how well they work in treating younger patients with Hodgkin lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To establish neurotoxicity of OEPA+COPP chemotherapy in young adults.

Secondary

* To determine response rates in patients treated with this regimen.
* To determine disease-free survival of patients treated with this regimen.
* To determine overall survival of patients treated with this regimen.
* To determine gonadal toxicity in patients treated with this regimen.

OUTLINE: Patients are assigned to treatment group according to stage.

* Group 1 (patients with stage 1A, 1B, or 2A disease): Patients receive OEPA chemotherapy comprising vincristine IV on days 1, 8, and 15; oral prednisolone on days 1-15; etoposide IV on days 1-5; and doxorubicin hydrochloride IV on days 1 and 15. Courses repeat every 28 days for 2 courses. Patients achieving a partial response also undergo radiotherapy after completion of chemotherapy; patients achieving a complete response do not undergo radiotherapy.
* Group 2 (patients with stage 2AE, 2B, or 3A disease): Patients receive 2 courses of OEPA chemotherapy as in group 1. Patients then receive COPP chemotherapy comprising cyclophosphamide IV on days 1 and 8; vincristine IV on days 1 and 8; oral procarbazine hydrochloride on days 1-15; and oral prednisolone on days 1-15. Courses repeat every 28 days for 2 courses. Patients also undergo radiotherapy after completion of chemotherapy.
* Group 3 (patients with stage 2BE, 3AE, 3BE, 3B, 4A, or 4B disease): Patients receive 2 courses of OEPA chemotherapy as in group 1. Patients then receive COPP chemotherapy as in group 2. Treatment with COPP chemotherapy repeats every 28 days for 4 courses. Patients also undergo radiotherapy after completion of chemotherapy.

In all groups, treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed periodically.

Peer Reviewed and Funded or Endorsed by Cancer Research UK.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Biopsy proven de-novo classical Hodgkin lymphoma

  * Any stage disease
  * No nodular lymphocyte-predominant Hodgkin lymphoma

PATIENT CHARACTERISTICS:

* No known or suspected HIV infection
* No pre-existing neurological disorder
* No serious comorbidity which may prevent administration of study treatment
* No other previous malignancy
* Not pregnant or nursing
* Fertile patients must use effective contraception during and for up to 1 year after completion of study treatment
* Creatinine ≤ 1.5 times upper limit of normal (ULN) unless due to the lymphoma
* ALT/AST ≤ 1.5 times ULN unless due to the lymphoma
* Bilirubin ≤ 2 times ULN unless due to the lymphoma

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy or radiotherapy
* No prior organ transplant

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2008-03; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Neurotoxicity due to the intensive use of Vinca alkaloids | End of treatment

SECONDARY OUTCOMES:
Response rate | End of treatment
Disease-free survival | Not specified in protocol
Overall survival | Not specified in protocol
Gonadal toxicity | Not specified in protocol

CONTACTS AND LOCATIONS:
Overall Officials: Kirit Ardeshna, Principal Investigator — University College London Hospitals
Locations (5):
- United Kingdom (5):
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - University College Hospital - London, London, England
  - King's College Hospital, London, England
  - Northern Centre for Cancer Treatment at Newcastle General Hospital, Newcastle upon Tyne, England
  - Mount Vernon Cancer Centre at Mount Vernon Hospital, Northwood, England